CLINICAL TRIAL: NCT01663792
Title: Dietary Seaweed and Early Breast Cancer: A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: DAMD-17-98-1-8207
Record Dates: First submitted 2012-08-09; First posted 2012-08-13 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Seaweed Associated Changes in Healthy Subjects
Keywords: urokinase receptor; protein expression; seaweed (Undaria pinnatifida)
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): 5 g/d placebo (maltodextrin)in 10 500-mg capsules for 1 month
  Interventions: Other: Placebo
- Seaweed (Experimental): Seaweed (Undaria pinnatifida) given orally in ten 500-mg capsules for 1 month
  Interventions: Other: Seaweed
- Placebo2 (Placebo Comparator): 5 g/d placebo in 10 500-mg capsules for one month
  Interventions: Other: Placebo2

INTERVENTIONS:
Other: Seaweed — Ten 500-mg capsules to be taken orally each day for 1 month
  Other Names: Undaria pinnatifida
  Arms: Seaweed
Other: Placebo — Ten 500-mg capsules to be taken orally each day for 1 month
  Other Names: Maltodextrin
  Arms: Placebo
Other: Placebo2 — Ten 500-mg capsules to be taken orally each day for 1 month
  Other Names: Maltodextrin
  Arms: Placebo2

SUMMARY:
Could daily consumption of seaweed help explain lower postmenopausal breast cancer (BC) incidence and mortality rates in Japan? This small proof of principle clinical trial was designed to test the idea that the same amount of seaweed normally eaten in Japan would induce metabolic changes when given to non-seaweed consuming healthy postmenopausal American women. The participants were given 10 capsules a day (about 1 tablespoon) for 3 months. During the first month the capsules contained placebo, the second month seaweed, and the third month placebo. We collected blood and urine samples after each treatment period and tested for changes in protein expression that might be related to consuming seaweed.

DETAILED DESCRIPTION:
The relationship between the relative breast cancer (BC) risk and seaweed intake among humans is only now unfolding. A small body of research, both in vivo and in vitro, suggests seaweed may be useful in BC prevention (Funahashi et al. 1999; Teas et al. 1984; Yamamoto et al. 1987) . Seaweeds are specifically used to treat tumors in Traditional Chinese Medicine and Japanese folk medicine. On a population level, those people for whom seaweed is a regular part of their diet, most notably in Japan, have dramatically lower rates of BC (Hebert et al. 1998; Hebert and Rosen 1996; Kodama et al. 1991).

Epidemiologic studies done in Japan in the 1980s, before Westernized diets were common, reported that Japanese women had 1/3 the rate of premenopausal BC and 1/9 the rate of postmenopausal BC (Ferlay et al. 2001; Reddy et al. 1980). Even today, BC incidence rates for women in Japan are 20/100,000 compared to the U.S. average of 118/100,000 (Statistics 2007) . Although genetic predisposition has been proposed, when rates among migrants from Japan to the US are compared, BC incidence almost doubles after 10 years of residence in the US (20/100,000 to 35/100,000) (Shimizu et al. 1991), increase with each successive generation (LeMarchand et al. 1985). Japanese-American women who develop BC have significantly better survival rates than other American ethnic groups (Kanemori and Prygrocki 2005; Pineda et al. 2001). On the other hand, Asian-American women over 50 years of age living in Los Angeles, especially Japanese-American women, have one of the most rapidly increasing BC incidence rates (Deapen et al. 2002). These data support the hypothesis that lifestyle changes and possibly gene-nutrient interactions are important in BC susceptibility.

Seaweed is a typical part of East-Asian diets, although consumption varies widely among individuals (Fukuda et al. 2007). Seaweeds have no land equivalents in terms of their specific components of fiber (alginate), primary carotenoid (fucoxanthin), sulfated polysaccharide (fucoidan and laminarin), and polyphenol defense compounds, each of which has been reported to have strong anti-cancer activity (Kotake-Nara et al. 2005; Koyanagi et al. 2003; Miao et al. 1999; Son et al. 2003).

Many in vivo and in vitro studies of dietary seaweed report decreased angiogenesis and increased apoptosis of tumor cells (Konishi et al. 2006; Koyanagi et al. 2003; Sekiya et al. 2005), inhibition of tumor cell adhesion and metastasis (Liu et al. 2005) and enhanced immune responses (Maruyama et al. 2003; Maruyama et al. 2006). Nishino and colleagues have investigated seaweed modulation of the urokinase plasminogen system (Nishino et al. 1999; Nishino et al. 2000). Based on the wide range of antitumor effects, we investigated the possibility that seaweed could affect uPAR concentrations in women who consume seaweed. The urokinase-type plasminogen activator (uPA), urokinase-type plasminogen activator receptor (uPAR, CD87), and its plasminogen inhibitors 1 and 2 are central to the maintenance of homeostasis, directly affecting the extracellular matrix (ECM), inflammation, tissue repair. Increased concentrations have been shown to be associated with more rapid cancer progression (Foekens et al. 2000). Urinary concentration of uPAR is highly correlated with urinary uPA concentrations, and both are correlated with tissue concentration (Foekens et al. 2000; Sier et al. 2004).When uPA/uPAR concentrations are increased, there is increased ECM degradation that allows cancer cells to migrate, leading to metastases. Urokinase is also used therapeutically to treat serious conditions involving blood clots. In clinical studies, tissue concentration of uPA is an independent prognostic predictor of BC progression (Ceccarelli et al. 2010; Look et al. 2002).

We therefore included evaluation of one part of the urokinase system, uPAR, in this study as a possible biomarker for seaweed activity that might be related to BC prevention.

To further assess whether a dietary seaweed intervention could alter protein expression in urine and serum in a non-seaweed consuming population of healthy postmenopausal women, we used surface enhanced laser desorption/ionization time of flight coupled with mass spectrometer (SELDI-TOF-MS). Proteomic analyses have been used to identify cancer biomarkers with high sensitivity and specificity, including those related to BC (Gast et al. 2008; Shimizu et al. 1991; van Winden et al. 2009). SELDI has also been shown to be sensitive enough to be used to identify changes in serum associated with the addition of a novel food (green tea) (Tsuneki et al. 2004).

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Postmenopausal (verified by follicle stimulating hormone (FSH) [23.0-116 mIU/ml]
* Omnivorous eating habits (including meat and dairy products more than twice per week)
* Limit alcoholic intake to ≤ 1 drink (12 g alcohol)/week

Exclusion Criteria:

* No allergies to seaweed, soy, shellfish or iodine
* No current use of tobacco
* No hormone replacement therapy
* For BC survivors, no chemotherapy or radiation treatments within the preceding 6 months
* No history of cancer (other than BC or squamous cell skin cancer) within the previous 20 years
* No current gastrointestinal disorders or diabetes
* No oral antibiotics taken in the previous 3 months

Ages: 45 Years to 68 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Urinary urokinase receptor concentration | 3 months
  ELISA test for uPAR concentration
Surface Enhanced Laser Desorption/Ionization-Time Of Flight-Mass Spectrometry (SELDI-TOF-MS)identification of urinary and serum protein changes | 3 months
  SELDI-TOF-MS was used to measure urinary and serum protein changes

SECONDARY OUTCOMES:
Urinary iodine concentrations | 3 months
  Urinary iodine concentration changes were used to indicate adherence to taking the seaweed supplement.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Teas, Ph.D., Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina Cancer Research Center, Columbia, South Carolina, United States

REFERENCES:
- [Background] Funahashi H, Imai T, Tanaka Y, Tsukamura K, Hayakawa Y, Kikumori T, Mase T, Itoh T, Nishikawa M, Hayashi H, Shibata A, Hibi Y, Takahashi M, Narita T. Wakame seaweed suppresses the proliferation of 7,12-dimethylbenz(a)-anthracene-induced mammary tumors in rats. Jpn J Cancer Res. 1999 Sep;90(9):922-7. doi: 10.1111/j.1349-7006.1999.tb00836.x. PMID 10551319
- [Background] Teas J, Harbison ML, Gelman RS. Dietary seaweed (Laminaria) and mammary carcinogenesis in rats. Cancer Res. 1984 Jul;44(7):2758-61. PMID 6426785
- [Background] Yamamoto I, Maruyama H, Moriguchi M. The effect of dietary seaweeds on 7,12-dimethyl-benz[a]anthracene-induced mammary tumorigenesis in rats. Cancer Lett. 1987 May;35(2):109-18. doi: 10.1016/0304-3835(87)90033-4. PMID 3107796
- [Background] Hebert JR, Rosen A. Nutritional, socioeconomic, and reproductive factors in relation to female breast cancer mortality: findings from a cross-national study. Cancer Detect Prev. 1996;20(3):234-44. PMID 8769718
- [Background] Kodama M, Kodama T, Miura S, Yoshida M. Nutrition and breast cancer risk in Japan. Anticancer Res. 1991 Mar-Apr;11(2):745-54. PMID 2064329
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Estimating the world cancer burden: Globocan 2000. Int J Cancer. 2001 Oct 15;94(2):153-6. doi: 10.1002/ijc.1440. No abstract available. PMID 11668491
- [Background] Reddy BS, Cohen LA, McCoy GD, Hill P, Weisburger JH, Wynder EL. Nutrition and its relationship to cancer. Adv Cancer Res. 1980;32:237-345. doi: 10.1016/s0065-230x(08)60363-2. No abstract available. PMID 6258405
- [Background] Shimizu H, Ross RK, Bernstein L, Yatani R, Henderson BE, Mack TM. Cancers of the prostate and breast among Japanese and white immigrants in Los Angeles County. Br J Cancer. 1991 Jun;63(6):963-6. doi: 10.1038/bjc.1991.210. PMID 2069852
- [Background] LeMarchand L, Kolonel LN, Nomura AM. Breast cancer survival among Hawaii Japanese and Caucasian women. Ten-year rates and survival by place of birth. Am J Epidemiol. 1985 Oct;122(4):571-8. doi: 10.1093/oxfordjournals.aje.a114136. PMID 4025300
- [Background] Kanemori M, Prygrocki M. Results of breast conservation therapy from a single-institution community hospital in Hawaii with a predominantly Japanese population. Int J Radiat Oncol Biol Phys. 2005 May 1;62(1):193-7. doi: 10.1016/j.ijrobp.2004.08.054. PMID 15850921
- [Background] Pineda MD, White E, Kristal AR, Taylor V. Asian breast cancer survival in the US: a comparison between Asian immigrants, US-born Asian Americans and Caucasians. Int J Epidemiol. 2001 Oct;30(5):976-82. doi: 10.1093/ije/30.5.976. PMID 11689507
- [Background] Deapen D, Liu L, Perkins C, Bernstein L, Ross RK. Rapidly rising breast cancer incidence rates among Asian-American women. Int J Cancer. 2002 Jun 10;99(5):747-50. doi: 10.1002/ijc.10415. PMID 12115511
- [Background] Fukuda S, Saito H, Nakaji S, Yamada M, Ebine N, Tsushima E, Oka E, Kumeta K, Tsukamoto T, Tokunaga S. Pattern of dietary fiber intake among the Japanese general population. Eur J Clin Nutr. 2007 Jan;61(1):99-103. doi: 10.1038/sj.ejcn.1602505. Epub 2006 Aug 2. PMID 16885928
- [Background] Kotake-Nara E, Asai A, Nagao A. Neoxanthin and fucoxanthin induce apoptosis in PC-3 human prostate cancer cells. Cancer Lett. 2005 Mar 18;220(1):75-84. doi: 10.1016/j.canlet.2004.07.048. PMID 15737690
- [Background] Koyanagi S, Tanigawa N, Nakagawa H, Soeda S, Shimeno H. Oversulfation of fucoidan enhances its anti-angiogenic and antitumor activities. Biochem Pharmacol. 2003 Jan 15;65(2):173-9. doi: 10.1016/s0006-2952(02)01478-8. PMID 12504793
- [Background] Miao HQ, Elkin M, Aingorn E, Ishai-Michaeli R, Stein CA, Vlodavsky I. Inhibition of heparanase activity and tumor metastasis by laminarin sulfate and synthetic phosphorothioate oligodeoxynucleotides. Int J Cancer. 1999 Oct 29;83(3):424-31. doi: 10.1002/(sici)1097-0215(19991029)83:33.0.co;2-l. PMID 10495437
- [Background] Son EW, Rhee DK, Pyo S. Antiviral and tumoricidal activities of alginate-stimulated macrophages are mediated by different mechanisms. Arch Pharm Res. 2003 Nov;26(11):960-6. doi: 10.1007/BF02980206. PMID 14661863
- [Background] Konishi I, Hosokawa M, Sashima T, Kobayashi H, Miyashita K. Halocynthiaxanthin and fucoxanthinol isolated from Halocynthia roretzi induce apoptosis in human leukemia, breast and colon cancer cells. Comp Biochem Physiol C Toxicol Pharmacol. 2006 Jan-Feb;142(1-2):53-9. doi: 10.1016/j.cbpc.2005.10.005. Epub 2005 Dec 7. PMID 16337836
- [Background] Sekiya M, Funahashi H, Tsukamura K, Imai T, Hayakawa A, Kiuchi T, Nakao A. Intracellular signaling in the induction of apoptosis in a human breast cancer cell line by water extract of Mekabu. Int J Clin Oncol. 2005 Apr;10(2):122-6. doi: 10.1007/s10147-004-0469-2. PMID 15864698
- [Background] Liu JM, Bignon J, Haroun-Bouhedja F, Bittoun P, Vassy J, Fermandjian S, Wdzieczak-Bakala J, Boisson-Vidal C. Inhibitory effect of fucoidan on the adhesion of adenocarcinoma cells to fibronectin. Anticancer Res. 2005 May-Jun;25(3B):2129-33. PMID 16158954
- [Background] Maruyama H, Tamauchi H, Iizuka M, Nakano T. The role of NK cells in antitumor activity of dietary fucoidan from Undaria pinnatifida sporophylls (Mekabu). Planta Med. 2006 Dec;72(15):1415-7. doi: 10.1055/s-2006-951703. Epub 2006 Oct 20. PMID 17054048
- [Background] Maruyama H, Tamauchi H, Hashimoto M, Nakano T. Antitumor activity and immune response of Mekabu fucoidan extracted from Sporophyll of Undaria pinnatifida. In Vivo. 2003 May-Jun;17(3):245-9. PMID 12929574
- [Background] Nishino T, Yamauchi T, Horie M, Nagumo T, Suzuki H. Effects of a fucoidan on the activation of plasminogen by u-PA and t-PA. Thromb Res. 2000 Sep 15;99(6):623-34. doi: 10.1016/s0049-3848(00)00289-9. PMID 10974349
- [Background] Nishino T, Fukuda A, Nagumo T, Fujihara M, Kaji E. Inhibition of the generation of thrombin and factor Xa by a fucoidan from the brown seaweed Ecklonia kurome. Thromb Res. 1999 Oct 1;96(1):37-49. doi: 10.1016/s0049-3848(99)00060-2. PMID 10554083
- [Background] Look MP, van Putten WL, Duffy MJ, Harbeck N, Christensen IJ, Thomssen C, Kates R, Spyratos F, Ferno M, Eppenberger-Castori S, Sweep CG, Ulm K, Peyrat JP, Martin PM, Magdelenat H, Brunner N, Duggan C, Lisboa BW, Bendahl PO, Quillien V, Daver A, Ricolleau G, Meijer-van Gelder ME, Manders P, Fiets WE, Blankenstein MA, Broet P, Romain S, Daxenbichler G, Windbichler G, Cufer T, Borstnar S, Kueng W, Beex LV, Klijn JG, O'Higgins N, Eppenberger U, Janicke F, Schmitt M, Foekens JA. Pooled analysis of prognostic impact of urokinase-type plasminogen activator and its inhibitor PAI-1 in 8377 breast cancer patients. J Natl Cancer Inst. 2002 Jan 16;94(2):116-28. doi: 10.1093/jnci/94.2.116. PMID 11792750
- [Background] Foekens JA, Peters HA, Look MP, Portengen H, Schmitt M, Kramer MD, Brunner N, Janicke F, Meijer-van Gelder ME, Henzen-Logmans SC, van Putten WL, Klijn JG. The urokinase system of plasminogen activation and prognosis in 2780 breast cancer patients. Cancer Res. 2000 Feb 1;60(3):636-43. PMID 10676647
- [Background] Boonstra MC, Verspaget HW, Ganesh S, Kubben FJ, Vahrmeijer AL, van de Velde CJ, Kuppen PJ, Quax PH, Sier CF. Clinical applications of the urokinase receptor (uPAR) for cancer patients. Curr Pharm Des. 2011;17(19):1890-910. doi: 10.2174/138161211796718233. PMID 21711239
- [Background] Ceccarelli F, Fuso A, Civitelli L, Ranieri E, Caprio G, Pagni P, Rengo M, Scarpa S. Urokinase expression in course of benign and malignant mammary lesions: comparison between nodular and healthy tissues. J Cancer Res Clin Oncol. 2010 Jan;136(1):157-63. doi: 10.1007/s00432-009-0694-1. Epub 2009 Oct 14. PMID 19826838
- [Background] Gast MC, Schellens JH, Beijnen JH. Clinical proteomics in breast cancer: a review. Breast Cancer Res Treat. 2009 Jul;116(1):17-29. doi: 10.1007/s10549-008-0263-3. Epub 2008 Dec 11. PMID 19082706
- [Background] van Winden AW, Gast MC, Beijnen JH, Rutgers EJ, Grobbee DE, Peeters PH, van Gils CH. Validation of previously identified serum biomarkers for breast cancer with SELDI-TOF MS: a case control study. BMC Med Genomics. 2009 Jan 19;2:4. doi: 10.1186/1755-8794-2-4. PMID 19152674
- [Background] Tsuneki H, Ishizuka M, Terasawa M, Wu JB, Sasaoka T, Kimura I. Effect of green tea on blood glucose levels and serum proteomic patterns in diabetic (db/db) mice and on glucose metabolism in healthy humans. BMC Pharmacol. 2004 Aug 26;4:18. doi: 10.1186/1471-2210-4-18. PMID 15331020